CLINICAL TRIAL: NCT04652505
Title: Coping With COVID: The Effect of the COVID-19 Public Health Crisis on Mental Well-Being in Cancer Patients Seen at the Psychiatric Oncology Clinic
Brief Title: Effect of the COVID-19 Public Health Crisis on the Mental Health and Physical Well-Being of Cancer Patients, the Coping With COVID Study
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0451; NCI-2020-06556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0451 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-11; First posted 2020-12-03 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — COVID-19; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires): Patients complete 3 questionnaires online over 15 minutes regarding coping strategies that may have been used, mental health and physical well-being in the past month, and if they have been following certain behaviors which the WHO has recommended during the coronavirus pandemic, such as regular hand washing and social distancing.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study determines how the threat of the coronavirus has affected the mental health and physical well-being of cancer patients seen at the psychiatric oncology clinic, and how they have coped with any related stress. Questionnaires that assess coping strategies and behaviors for decreasing disease transmission may help researchers create recommendations for future public health crises and pandemics.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine how the coronavirus disease 2019 (COVID-19) public health crisis affected mental well-being in cancer patients seen at the psychiatric oncology clinic.

SECONDARY OBJECTIVES:

I. To determine how the COVID-19 public health crisis affected physical well-being and substance use in cancer patients seen at the psychiatric oncology clinic.

II. To determine how patient coping strategies and levels of apathy affected mental and physical health symptoms and substance use during COVID-19 in patients seen at the psychiatric oncology clinic.

III. To determine the association of coping strategies and levels of apathy with proclivity to engage in health behaviors intended to decrease the transmission of the disease during the COVID-19 pandemic in patients seen at the psychiatric oncology clinic.

OUTLINE:

Patients complete 3 questionnaires online over 15 minutes regarding coping strategies that may have been used, mental health and physical well-being in the past month, and if they have been following certain behaviors which the World Health Organization (WHO) has recommended during the coronavirus pandemic, such as regular hand washing and social distancing.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients seen by providers of the psychiatric oncology clinic at least once between November 1, 2019 and February 29, 2020 and at least once between April 10, 2020 and June 10, 2020
* Speaking English as indicated in their medical chart

Exclusion Criteria:

* Patients who are pregnant as recorded in their medical chart
* Incarcerated
* With a recorded diagnosis of a formal thought disorder
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who received care at the psychiatric oncology clinic during the COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Patient-reported severity of depression | Baseline
  sum score on the Patient Health Questionnaire, a 9-item scale with a sumscore ranging between 0 and 27, with a higher score indicating more-severe depression.
Patient-reported severity of anxiety | Baseline
  sum score on the generalized anxiety disorder questionnaire, a 7-item scale with sumscore range between 0 and 21. A higher score indicates higher severity of anxiety.
Patient-reported severity of distress | Baseline
  score on the National Comprehensive Cancer Network Distress Thermometer, a one-item 0-10 scale. A higher score indicates higher distress.

SECONDARY OUTCOMES:
Patient-reported physical symptoms | Baseline
  Physical symptoms are assessed with individual-item response on the Edmonton Symptom Assessment Scale by the clinic. The ESAS includes 6 somatic symptom items, each of which is to be rated on a 0-10 scale, with higher scores indicating higher severity of the symptom.
Substance use | Baseline
  Substance use is documented by the treating physician and will be abstracted from clinic notes.
Patient-reported coping strategy | Baseline
  Assessed using the brief COPE questionnaire. Will examine active versus avoidant coping. Active coping, planning, positive reframing, acceptance, humor, religion, emotional support-seeking, and instrumental support-seeking will be considered active coping strategies. Self-distraction, denial, venting, substance use, behavioral disengagement, and self-blame will be considered maladaptive coping strategies.
Patient-reported levels of apathy | Baseline
  The Apathy evaluation Scale is an 18-item scale with a sum score ranging between 18 and 72. A higher scores indicates higher apathy..
Patient-reported engagement in the 5 health behaviors endorsed by World Health Organization intended to curb the spread of the coronavirus | Baseline
  Patients indicate how often during the pandemic they engaged in the following 5 behaviors endorsed by the World Health Organization to decrease the transmission of coronavirus disease 2019 (COVID-19): washing hands regularly for 20 seconds with soap and water or alcohol-based hand rub, covering nose and mouth with a disposable tissue or flexed elbow when you cough or sneeze, avoiding close contact with people who are unwell, staying home and self-isolating from others in the household when feeling unwell, avoiding touching eyes, nose, and mouth when hands are unclean. The behaviors will be assessed on a Likert scale of 1-5, with 1 being "never" and 5 being "always". A not available (N/A) option will be given for staying home and self-isolating from others when feeling unwell, since participants may not experience a period of feeling unwell.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara E Lacourt, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org